CLINICAL TRIAL: NCT03244618
Title: A Medical Device Study to Measure the Efficacy of a Toothpaste Containing Calcium-silicate/Phosphate on Dentinal Hypersensitivity Compared to a Control Toothpaste Containing Fluoride.
Brief Title: A Study to Measure the Efficacy of a Toothpaste on Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORL-SEN-2530
Record Dates: First submitted 2017-07-18; First posted 2017-08-09 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSSP Toothpaste (Experimental): Toothpaste containing Calcium Silicate and Sodium Phosphate
  Interventions: Device: CSSP Toothpaste
- Fluoride Toothpaste (Placebo Comparator): Toothpaste containing Sodium monofluorphosphate
  Interventions: Device: Fluoride Toothpaste

INTERVENTIONS:
Device: CSSP Toothpaste — Toothpaste containing calcium silicate, sodium phosphate and sodium monofluorophosphate
  Arms: CSSP Toothpaste
Device: Fluoride Toothpaste — Toothpaste containing sodium monofluorphosphate
  Arms: Fluoride Toothpaste

SUMMARY:
Double blind parallel study to measure the efficacy of a toothpaste containing calcium-silicate/phosphate on dentinal hypersensitivity compared to a control toothpaste containing fluoride

DETAILED DESCRIPTION:
This is a double blind parallel design, with respect to the clinical assessor and subject, study. A minimum of 280 (140 per group), male and female subjects will be recruited to ensure that a minimum of 200 subjects (100 per group) complete the study. Subjects will attend the test site on six (6) occasions.

Subjects will be screened according to the inclusion and exclusion criteria. Suitable subjects will be given a standard fluoride toothpaste and a toothbrush to use for the following four to six weeks (Run-in Phase).

On completion of the run in phase, the subjects will have a baseline sensitivity and soft tissue assessments conducted and randomised to product (visit 3).

Subjects will be randomly assigned to the test groups.

Subjects will be given sufficient supplies of their allocated toothpaste and a toothbrush to use for the following 2 weeks. Instructions for use (IFUs) will be given to the subjects along with a toothbrushing diary and an appointment to return to the test site 2 weeks (+/-1 day) later.

At the Day 14 visit, subjects will have the dentinal hypersensitivity and soft tissue assessments repeated.

Subjects will be given sufficient supplies of their allocated toothpaste and a toothbrush to use for the following 2 weeks. A fresh toothbrushing diary will be given to the subject along with an appointment to return to the test site 2 weeks later (Week 4 assessment). Subjects will be instructed to brush their teeth as per the IFU for the following 2 weeks.

At the Day 28 visit subjects will have the dentinal hypersensitivity and soft tissue assessments repeated. Prior to leaving the study site, the subjects will be asked to brush their teeth as per the IFU. Subjects will be requested to brush their teeth at a specific time and return to the study site the following day.

At the Day 29 visit, subjects will have the dentinal hypersensitivity and soft tissue assessments repeated. On completion of the assessments, subjects will receive their remuneration for the participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 years and older.
* Willing and physically able to carry out all study procedures.
* Willing and able to give written informed consent and complete a medical history form.
* Have at least one hypersensitive tooth in two quadrants, which are anterior to the molars and demonstrate cervical dentine, which have an air-blast hypersensitivity score of 2 or 3 on the Schiff sensitivity scale at Screening and Baseline and a tactile hypersensitivity score of 10-20 grams of force at baseline.
* Willing to comply with the oral hygiene and food and drink restrictions.

Exclusion Criteria:

* Subjects who have used anti sensitivity products in the 4 weeks prior to screening
* Subjects with an active oral ulcer (Aphthous ulcer), or have similar experience within past 1 month.
* Subjects who use a powered toothbrush at least 4 times a week to brush their teeth
* Subjects whose indicator teeth have abnormal oral pathology, for example:

  * Extensive restorations.
  * Observable caries.
  * Observable cracked enamel.
  * Leaking fillings or other restorations.
  * Cracked Tooth Syndrome
  * Suspected pulp pathology/abscess/pulpitis.
  * Atypical facial pain
  * Any tooth surface adjacent to those surfaces under investigation, which in the opinion of the investigator have any other condition(s) that provide confusing symptoms to those of cervical dentine hypersensitivity.
* Currently undergoing dental treatment, including orthodontic treatment.
* Subjects who have had vital bleaching within 4 weeks of the screening visit
* Known allergies to any toothpaste ingredients, including the flavour components.
* Obvious physical disability reducing tooth brushing ability.
* Receiving concomitant medication/therapy that might affect dentine hypersensitivity, e.g. regular use of analgesics, anti-histamines, non-steroidal anti-inflammatory drug and selective serotonin reuptake inhibitor medication
* Severe gingivitis, periodontitis and/or marked tooth mobility.
* Gingival surgery in the previous six months.
* In the opinion of the investigator unable to comply fully with the trial requirements.
* Participation in other dental clinical trials in the previous 28 days
* Subjects who have participated in an dentinal hypersensitivity study within the previous 1 month.
* Diabetic (both Type 1 and Type 2)
* Medical condition(s) and/or regular use of any medication, which either could affect the scientific validity of the study or if the subject was to participate in the study could, affect their wellbeing.
* Smokers or e-cigarette use or those who have smoked/vaped in the previous 12 months
* Brushing < 10 times a week during the Run-In period (self-reported)
* Using <17g or > 53g of toothpaste in a two week period during the test phase
* The subject is an employee of Unilever or the site conducting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola X West, Professor, Principal Investigator — University of Bristol
Locations (1):
- School of Oral and Dental Science, Bristol, United Kingdom

REFERENCES:
- [Derived] Seong J, Newcombe RG, Matheson JR, Weddell L, Edwards M, West NX. A randomised controlled trial investigating efficacy of a novel toothpaste containing calcium silicate and sodium phosphate in dentine hypersensitivity pain reduction compared to a fluoride control toothpaste. J Dent. 2020 Jul;98:103320. doi: 10.1016/j.jdent.2020.103320. Epub 2020 Jun 1. PMID 32497553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single center in Bristol, United Kingdom.
Pre-assignment Details: Participants brushed for 4-6 weeks with fluoride toothpaste during run-in period between enrollment and randomization. 272 participants were enrolled out of which 263 were randomized. Reasons for participant not being randomized:
  * Did not meet Baseline inclusion criteria (n=1)
  * Withdrawal by subject (n=6)
  * Lost to follow-up (n=2)
Groups:
- CSSP Toothpaste: Toothpaste containing calcium silicate, sodium phosphate and sodium monofluorophosphate. Participants were asked to brush for two minutes with the toothpaste twice per day, morning and evening, using their normal routine. After the evening brush, partipants were instructed to massage a pea sized amount of the toothpaste into the sensitive surfaces of the two selected sensitive teeth for 30 seconds.
- Fluoride Toothpaste: Toothpaste containing sodium monofluorphosphate. Participants were asked to brush for two minutes with the toothpaste twice per day, morning and evening, using their normal routine. After the evening brush, partipants were instructed to massage a pea sized amount of the toothpaste into the sensitive surfaces of the two selected sensitive teeth for 30 seconds.
Period: Overall Study
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
Started | 132 | 131
Week 2 | 128 | 125
Completed | 125 | 122
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 3 | 4
Not completed — Protocol Violation | 4 | 3
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste | Total
Number analyzed (Participants) | 132 | 131 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (12.7) | 37.4 (13.5) | 35.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 143
  Male | 60 | 60 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 106 | 104 | 210
  Asian | 13 | 16 | 29
  Black | 10 | 11 | 21
  Other | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 132 | 131 | 263
Thermo-evaporative (Schiff air blast) stimuli [Mean (Standard Deviation); unit: units on a scale] — Air blast sensitivity assessed by directing a one-second blast of air onto the exposed buccal root surface of sensitive tooth. Sensitivity recorded: 0 = Tooth/Subject does not respond; 1 Tooth/subject responds but does not request discontinuation; 2 Tooth/subject responds and requests discontinuation or moves;3 Tooth/subject responds, considers stimulus to be painful, and requests discontinuation. Each subject will be characterised at each visit by the average of the relevant scores for the two indicator teeth. HIgher score is worse outcome.
  units on a scale | 2.193 (0.336) | 2.256 (0.336) | 2.224 (0.337)

OUTCOME MEASURES:

1. Primary Outcome: Thermo-evaporative (Schiff Air Blast) Stimuli
Description: Air blast sensitivity assessed by directing a one-second blast of air onto the exposed buccal root surface of sensitive tooth. Sensitivity recorded: 0 = Tooth/Subject does not respond; 1 Tooth/subject responds but does not request discontinuation; 2 Tooth/subject responds and requests discontinuation or moves;3 Tooth/subject responds, considers stimulus to be painful, and requests discontinuation. Each subject will be characterised at each visit by the average of the relevant scores for the two indicator teeth. HIgher score is worse outcome.
Time Frame: 4-weeks of product use (Day 28)
Population: Analysis was based on all available data at week 4 from subjects who were randomised
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 125 | 122
score on a scale
  Baseline | 2.188 (0.334) | 2.246 (0.329)
  Week 4 | 1.268 (0.723) | 1.811 (0.624)
Statistical Analysis 1: Comparison: CSSP Toothpaste vs Fluoride Toothpaste; Test type: Superiority; p < 0.001, ANOVA; ANOVA model had treatment and gender as factors; Mean Difference (Final Values) = -0.544, 95% CI 2-sided [-0.712 to -0.377] — Difference is first named toothpaste minus second named toothpaste such that a negative difference favours first named toothpaste

2. Secondary Outcome: Tactile (Yeaple Probe) Stimuli
Description: The Yeaple score is recorded in terms of quantified reproducible force (range 10-60 grams with higher values indicating a better outcome). The Yeaple probe tip with a force of 10 grams is passed over the exposed dentin on the buccal surface of the selected teeth, apical to the cementenamel junction and the applied force in increased each time by 10 grams until the participant indicates that he/she is experiencing discomfort, or until 20 grams (baseline) or 60 grams (post product use) of force is reached. A higher value indicates lower levels of dentinal hypersensitivity. Each subject will be characterised at each visit by the average of the relevant scores for the two indicator teeth.
Time Frame: 4-weeks of product use (Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 125 | 122
score on a scale
  Baseline | 17.5 (3.46) | 16.6 (3.75)
  Week 4 | 38.2 (14.4) | 27.5 (11.7)
Statistical Analysis 1: Comparison: CSSP Toothpaste vs Fluoride Toothpaste; Test type: Superiority; p < 0.001, ANOVA; ANOVA model had treatment and gender as factors; Mean Difference (Final Values) = 10.8, 95% CI 2-sided [7.5 to 14.0] — Difference is first names toothpaste minus second named toothpaste such that a positive difference favours the first named toothpaste

3. Secondary Outcome: Visual Analogue Scale
Description: Visual Analogue Scale values were recorded to give the outcome variable per subject at the same time asSchiff assessment. The VAS values were assigned a numerical value in the conventional order from 0 (no pain) to 100 (extremely pain).
Time Frame: 4-weeks of product use (Day 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 125 | 122
score on a scale
  Baseline | 48.1 (20.5) | 49.9 (19.8)
  Week 4 | 31.1 (22.8) | 42.0 (22.1)
Statistical Analysis 1: Comparison: CSSP Toothpaste vs Fluoride Toothpaste; Test type: Superiority; p < 0.001, ANOVA; ANOVA model had treatment and gender as factors; Mean Difference (Final Values) = -11.0, 95% CI 2-sided [-16.4 to -5.5] — Difference is first named toothpaste minus second named toothpaste such that a negative difference favours the first named toothpaste

4. Other Pre Specified Outcome: Thermo-evaporative (Schiff Air Blast) Stimuli
Description: Air blast sensitivity assessed by directing a one-second blast of air onto the exposed buccal root surface of sensitive tooth. Sensitivity will be recorded: 0 = Tooth/Subject does not respond; 1 Tooth/subject responds but does not request discontinuation; 2 Tooth/subject responds and requests discontinuation or moves;3 Tooth/subject responds, considers stimulus to be painful, and requests discontinuation. Each subject will be characterised at each visit by the average of the relevant scores for the two indicator teeth.
Time Frame: Day 29, 12 hours after product use has ceased
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 125 | 122
score on a scale
  Baseline | 2.188 (0.334) | 2.246 (0.329)
  Day 29, 12hr after last product use | 1.044 (0.773) | 1.713 (0.671)
Statistical Analysis 1: Comparison: CSSP Toothpaste vs Fluoride Toothpaste; Test type: Superiority; p < 0.001, ANOVA; ANOVA model had treatment and gender as factors; Mean Difference (Final Values) = -0.670, 95% CI 2-sided [-0.850 to -0.489] — Difference is first named toothpaste minus second named toothpaste such that a negative value favours the first named toothpaste

5. Other Pre Specified Outcome: Tactile (Yeaple Probe) Stimuli
Description: as for outcome 2
Time Frame: Day 29, 12 hours after product use has ceased
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 125 | 122
score on a scale
  Baseline | 17.5 (3.46) | 16.6 (3.75)
  Day 29, 12hr after last product use | 41.5 (14.2) | 29.7 (11.9)
Statistical Analysis 1: Comparison: CSSP Toothpaste vs Fluoride Toothpaste; Test type: Superiority; p < 0.001, ANOVA; ANOVA model had treatment and gender as factors; Mean Difference (Final Values) = 11.9, 95% CI 2-sided [8.6 to 15.1] — Difference is first named toothpaste minus second named toothpaste such that a positive difference favours first named toothpaste

6. Other Pre Specified Outcome: Visual Analogue Scale
Description: Visual Analogue Scale values of the same teeth will be also be recorded to give the outcome variable per subject at the same time of Schiff assessment. The VAS values will be assigned a numerical value in the conventional order from 0 (no pain) to 100 (extremely pain).
Time Frame: Day 29, 12 hours after product use has ceased
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
Number analyzed (Participants) | 125 | 122
score on a scale
  Baseline | 48.1 (20.5) | 49.9 (19.8)
  Day 29, 12hr after last product use | 27.2 (23.2) | 38.1 (22.7)
Statistical Analysis 1: Comparison: CSSP Toothpaste vs Fluoride Toothpaste; Test type: Superiority; p < 0.001, ANOVA; ANOVA model had treatment and gender as factors; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-16.6 to -5.2] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From start of screening until final assessment visit (up to 61 days)
Description: Systematic assessment undertaken of oral soft tissues at assessment visits. Non-systematic assessment also used i.e. subject self-report.
Arm/Group | CSSP Toothpaste | Fluoride Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/131
Other Adverse Events (participants affected / at risk) | 2/132 | 4/131
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSSP Toothpaste (N=132) | Fluoride Toothpaste (N=131)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Cold (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03244618/Prot_SAP_000.pdf